CLINICAL TRIAL: NCT05533554
Title: Brief Intervention Based on the Theory of Planned Behavior to Reduce Alcohol Consumption in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Romero Reyes (Other)
Collaborators: Universidad Nacional de Educación a Distancia (Other)
Responsible Party: Sponsor-Investigator, Daniela Romero Reyes, Principal investigator, Universidad Autónoma de Tamaulipas
Organization: Universidad Autónoma de Tamaulipas (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 117
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Alcohol; Harmful Use
Keywords: Brief online intervention; Planned Behavior Theory; Hazardous and harmful use of alcohol; University Students
MeSH Terms: interventions — Ethanol; Economics

STUDY DESIGN:
Intervention Model Description: Experimental methodology with experimental group and control group on waiting list.
Who Masked: Participant, Outcomes Assessor
Masking Description: Simple, dynamic randomization will be carried out, balancing the groups based on sex (Female/Male). The masking will be single blind, where the researcher will know which participants will make up each group, said information will not be known to the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group with intervention (Experimental): The experimental group will receive the intervention. First, the group will undergo a pre-intervention evaluation lasting 120 minutes. The intervention will consist of two synchronized virtual sessions of brief intervention with a cognitive-behavioral approach where various persuasive communication strategies will be implemented, definition of hazardous alcohol consumption, establishment of a consumption goal, social skills to deal with pressure to consume and plan of pleasant activities alternative to consumption, each session will last 120 minutes. Four weeks after the end of the intervention, the experimental group will carry out the post-intervention evaluation session in a virtual synchronized manner with a duration of 120 minutes.
  Interventions: Behavioral: Brief Intervention Based on the Theory of Planned Behavior to Reduce Alcohol Consumption in University Students
- Control group (No Intervention): The control group will participate in a pre-intervention evaluation session. Four weeks after the end of the last intra-session evaluation session, the control group will participate in the post-intervention evaluation in a virtual synchronized manner with a duration of 120 minutes.

INTERVENTIONS:
Behavioral: Brief Intervention Based on the Theory of Planned Behavior to Reduce Alcohol Consumption in University Students — Cognitive-behavioral intervention where the key concepts of the Theory of Planned Behavior were operationalized from which two intervention sessions were formed and the most appropriate techniques were chosen to influence the key concepts of the theory: behavioral beliefs, subjective norms, perceived behavioral control and self-efficacy. The program is made up of 3 evaluation sessions (pre and post a month later) and 2 intervention sessions with a duration of 120 minutes each.
  Arms: Experimental group with intervention

SUMMARY:
Brief behavioral intervention designed from the guidelines of the Theory of Planned Action (TAP) of Ajzen (1991). It has the general objective of reducing the intention and hazardous and harmful consumption of alcohol in young university students in the first year of their undergraduate degree. The following specific objectives are considered: (a) Impact on the personal and descriptive norm by modifying the perception of the actual use of alcohol and its level of acceptance among the population of university students. (b) Modify attitudes towards consumption by reducing the value attributed to the expectations associated with risky alcohol consumption. (c) Increase perceived behavioral control and self-efficacy to avoid alcohol consumption behavior by: establishing a goal, consumption planning, and increase assertive communication.(d) Reduce the negative consequences of the use of alcohol in different situations of young people through pleasant healthy activities. e) Increase the intention to seek help for alcohol-related problems.The intervention will be developed through 3 phases. The first phase corresponds to the pre-intervention evaluation, the second phase concerns the two intervention sessions and the third phase is the post-intervention evaluation. Hypothesis: The mean alcohol consumption will be lower in young adults with hazardous and harmful alcohol consumption in the experimental group who received a brief online intervention compared to the control group.

DETAILED DESCRIPTION:
The hazardous and harmful consumption of alcohol in university students is a public health problem, as shown by various international studies. The consequences of consumption, the harmful effects of alcohol, impact various areas of the lives of young adults and those close to them, among which can be mentioned the increased risk of physical harm, legal problems, breach of school, relational responsibilities, negative social interactions, and processing can also be affected cognitive.

The WHO's report of Independent High-Level Commission on Noncommunicable Diseases states that national governments and cities should participate in measures related to noncommunicable diseases, including discouraging the harmful use of alcohol and promote mental health. The global strategy to reduce the harmful use of alcohol includes support for screening and preventive interventions related to hazardous alcohol use in primary health care and other settings. In Mexico, the General Health Law in its article 185, establishes the program for the prevention, reduction, and treatment of the harmful use of alcohol, attention to alcoholism, the prevention of diseases derived from it. Among its actions is the promotion of prevention, early detection, guidance, care, referral and treatment services for people and groups with harmful use of alcohol, avoiding all forms of stigmatization. The Official Mexican Standard 028 for the prevention, treatment, and control of addictions, refers to prevention as those actions aimed at reducing the non-therapeutic consumption of psychoactive substances and indicates that preventive programs must have a theoretical and methodological framework; include vulnerable populations, considering mainly the youth population.

From the international and national scene, the need to preventively attend to the harmful consumption of alcohol is evident, emphasizing the youth population. As measures in such circumstances, online interventions have been effective in reducing risky alcohol consumption, the Anglo-Saxon scientific literature supports the use of the Internet to carry out interventions aimed at reducing alcohol consumption in university students. In Latin America, a first systematic review on brief interventions reported that the interventions studied were given in a traditional face-to-face format, most of them in Brazil and Mexico, with heterogeneous theoretical and methodological approaches used, however, using the internet as a means to carry out brief interventions can be beneficial for university students who are in regions where there is little information on alcohol consumption or for students who have difficulties participating in face-to-face strategies, the brief interventions can serve as health literacy tools mental health that encourage young people to seek early help.

There is increasing evidence that public health interventions based on theories of social and behavioral sciences are more effective than those that do not have such a theoretical basis, the theory is a fundamental element of behavioral interventions, theories explain the pathways that lead or predict behavior and thus provide guidance on how to influence or modify said behavior.

The Theory of Planned Action is a strong theoretical basis for developing interventions to make changes in health-related behaviors. According to TAP, behavior is preceded by intentions, which in turn are shaped by attitudes, subjective norm, and perceived behavioral control. Attitudes are made up of behavioral beliefs (beliefs about the results of behavior and the evaluation of these results), the subjective norm is made up of normative beliefs, that is, beliefs about the normative expectations of others and the motivation to comply with them. these expectations, perceived behavioral control is integrated from control beliefs (beliefs about the presence of factors that can facilitate or hinder behavior), the perceived behavioral control construct is compatible with Bandura's perceived self-efficacy , which refers to the perception of confidence in being able to carry out a behavior, beliefs of self-efficacy or perceived behavioral control are located by TAP in a framework of relationships between attitudes, beliefs, intentions and behavior.

Study Design:

An experimental methodology is contemplated with an experimental group and a control group on a waiting list, with pre and post evaluation.

Population, sampling and sample:

The population will be made up of university students. The participants will be first-year university students. Through the G Power program, it is considered that for an effect size of .80, with a significance level of 0.05 and .80 power, each group (control and experimental) should be made up of 26 participants, 52 participants in total.

Procedure for data collection:

Quality assurance plan. In accordance with the Good Clinical Practices: Document of the Americas, procedures were developed for each of the four phases of the study

ELIGIBILITY:
Inclusion Criteria:

* Be a university student in the first or second year.
* Be between 18 and 29 years old.
* Voluntarily participate in the study.

Exclusion Criteria (post-hoc):

* Presence of severe mental disorder (e.g., psychotic disorders).
* Not having stable housing.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Mean change in score on the Alcohol Use Disorders Identification Questionnaire - Concise (AUDIT-C) | 4 weeks
  The AUDIT-C has 3 questions and is scored on a scale of 0 to 12. Each AUDIT-C question has 5 response options valued from 0 points to 4 points. Lower scores indicate a positive response to the intervention. The instrument will be applied in the preevaluation and up to four weeks after the end of the intervention.
Mean change in the amount of standard drinks ingested evaluated with the LIBARE Retrospective Baseline, from the initial evaluation, in two intra-sessions and two weeks after the end of the intervention | 4 weeks
  Instrument in the form of a calendar where the participant will be asked to record the days of consumption and the amount consumed according to the standard drink measure in a period of three months prior to the intervention. Afterwards, four weeks post-intervention, the participant will be asked to fill out this calendar for the 30 days that have elapsed since the last session. Fewer days of consumption, less number of drinks per consumption occasion and number of standard drinks ingested indicate a positive response to the intervention.

SECONDARY OUTCOMES:
Mean change in the assessment of the consequences of consumption (behavioral beliefs: attitude) measured through the TAP Questionnaire for alcohol consumption | 4 weeks
  Subscale made up of 25 items that evaluate attitude through consequences of consumption highly valued in the study population (behavioral beliefs), with 5 response options scored from 0 to 4 from "not important at all" to "very important". Lower scores indicate a positive response to the intervention. Participants will be asked to answer the instrument one day before and one day after the intervention and four weeks after it.
Mean change in subjective, personal and descriptive norms measured through the TAP Questionnaire for alcohol consumption | 4 weeks
  Subscale composed of 2 items of subjective norms and 1 item of descriptive norms, with 5 Likert-type response options scored from 0 to 4, lower scores indicate a positive response to the intervention. It also includes 1 personal norm item with 5 response options scored from 0 to 4; higher scores on this item indicate a positive response to the intervention. Participants will be asked to answer the instrument one day before and one day after the intervention and four weeks after it.
Mean change in perceived behavioral control measured through the TAP Questionnaire for alcohol consumption | 4 weeks
  Subscale composed of 2 items of perceived behavioral control towards alcohol consumption, scored from 0 to 4, lower scores on these items indicate a positive response to the intervention. The scale is also integrated by 3 items of perceived behavioral control towards alcohol abstinence, scored from 0 to 4, higher scores in these items indicate a positive response to the intervention. Participants will be asked to answer the instrument one day before and one day after the intervention and four weeks after it.
Mean change in the intention to consume alcohol measured through the TAP Questionnaire for alcohol consumption | 4 weeks
  Scale composed of 3 items of alcohol consumption intention with five response options from 0 to 4. Lower scores indicate a positive response to the intervention. Participants will be asked to answer the instrument one day before and one day after the intervention and four weeks after it.
Mean change in the degree of self-efficacy to face situations of alcohol consumption measured through the Brief Situational Confidence Questionnaire for university students | 4 weeks
  The objective of this scale is to measure the concept of self-efficacy in relation to the participant's perception of their ability to deal effectively with situations of alcohol consumption. The scale is made up of a single dimension of 4 items with response options from 0 (I do not trust myself) to 3 (I totally trust myself), the higher the score, the higher the self-efficacy. Higher scores on this scale indicate a positive response to the intervention. Participants will be asked to answer the instrument one day before and one day after the intervention and four weeks after it.
Measurement of adverse events through the implementation of the Scale on Consequences of Alcohol Consumption in University Students | 4 weeks
  This instrument measures consequences of alcohol consumption. It has 25 items with "yes/no" response options for the occurrence of consequences and for the frequency of occurrence of consequences in the last month: 0 times, 1 time, 2 times, 3 times, 4 to 5 times, 6 to 7 times, 12 to 20 months, more than 21 times. Fewer number and frequency of consequences indicate a positive response to the intervention. Participants will be asked to answer the instrument one day before the intervention and four weeks after it.
Help-seeking intention in young adults with hazardous and harmful alcohol consumption questionnaire (IH-RHAC) | 4 weeks
  instrument aims to measure help-seeking intention and attitude, subjective norm, and perceived behavioral control (operationalized as self-efficacy) based on the beliefs underlying these constructs: behavioral beliefs, normative beliefs, respectively, including the variable seeking help in the past. The scale is composed of five sections: (a) attitude, (b) subjective norm, (c) self-efficacy, (d) help-seeking intentions, and (e) past help-seeking. Responses were scored on a Likert-type scale from 1 to 5. Participants will be asked to answer the instrument one day before and one day after the intervention and four weeks after it.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Romero Reyes, Psychology, Principal Investigator — Universidad Autónoma de Tamaulipas; Juan Antonio Moriano León, Psychology, Study Director — Universidad Nacional de Educación a Distancia; José Luis Ybarra Sagarduy, Psychology, Study Director — Universidad Autónoma de Tamaulipas
Locations (1):
- Universidad Autónoma de Tamaulipas, Victoria, Tamaulipas, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data will be available to researchers who request it by email to danielaromeroreyes@gmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years
Access Criteria: Previous request to Daniela Romero Reyes (danielaromeroreyes@gmail.com)

REFERENCES:
- [Background] Ajzen I. The theory of planned behavior. Organizational behavior and human decision processes. 1991;50(2):179-211.
- [Background] Davoren MP, Demant J, Shiely F, Perry IJ. Alcohol consumption among university students in Ireland and the United Kingdom from 2002 to 2014: a systematic review. BMC Public Health. 2016 Feb 19;16:173. doi: 10.1186/s12889-016-2843-1. PMID 26895824
- [Background] Krieger H, Young CM, Anthenien AM, Neighbors C. The Epidemiology of Binge Drinking Among College-Age Individuals in the United States. Alcohol Res. 2018;39(1):23-30. doi: 10.35946/arcr.v39.1.05. PMID 30557145
- [Background] Yi S, Ngin C, Peltzer K, Pengpid S. Health and behavioral factors associated with binge drinking among university students in nine ASEAN countries. Subst Abuse Treat Prev Policy. 2017 Jun 26;12(1):32. doi: 10.1186/s13011-017-0117-2. PMID 28651601
- [Background] Bhochhibhoya A, Hayes L, Branscum P, Taylor L. The Use of the Internet for Prevention of Binge Drinking Among the College Population: A Systematic Review of Evidence. Alcohol Alcohol. 2015 Sep;50(5):526-35. doi: 10.1093/alcalc/agv047. Epub 2015 Jun 4. PMID 26047832
- [Background] Mota R, Fuentes-Mejía C, Belchior M, Pinto G, León F, Cruvinel E. Brief interventions for substance abuse in Latin America: a systematic review. Psychology in Study. 2019;(24).
- [Background] Tebb KP, Erenrich RK, Jasik CB, Berna MS, Lester JC, Ozer EM. Use of theory in computer-based interventions to reduce alcohol use among adolescents and young adults: a systematic review. BMC Public Health. 2016 Jun 17;16:517. doi: 10.1186/s12889-016-3183-x. PMID 27317330
- [Background] Glanz K, Bishop DB. The role of behavioral science theory in development and implementation of public health interventions. Annu Rev Public Health. 2010;31:399-418. doi: 10.1146/annurev.publhealth.012809.103604. PMID 20070207
- [Background] Norman P, Cameron D, Epton T, Webb TL, Harris PR, Millings A, Sheeran P. A randomized controlled trial of a brief online intervention to reduce alcohol consumption in new university students: Combining self-affirmation, theory of planned behaviour messages, and implementation intentions. Br J Health Psychol. 2018 Feb;23(1):108-127. doi: 10.1111/bjhp.12277. Epub 2017 Sep 20. PMID 28941040
- [Background] Ajzen I. Design and evaluation guided by the theory of planned behavior. Soc psychol Eval, Guilford Publications. 2011:74-100.
- [Background] Hurlbut SC, Sher KJ. Assessing alcohol problems in college students. J Am Coll Health. 1992 Sep;41(2):49-58. doi: 10.1080/07448481.1992.10392818. PMID 1460173
- [Background] Salazar GM, Muro MD, Udave MA, Leos FM. Adaptation of the Young Adult Alcohol Problem Screening Test (YAAPST) with university students from Mexico. Research and science. 2012;20(56):44-52.
- See also: World Health Organization. (2018) Report of the WHO Independent High-Level Commission on Noncommunicable Diseases. Geneva, Switzerland. — https://apps.who.int/iris/handle/10665/272712
- See also: Chamber of Deputies of the H. Congress of the Union. (2022, May 16) General Health Law. Official Journal of the Federation. — https://www.diputados.gob.mx/LeyesBiblio/ref/lgs/LGS_ref131_16may22.pdf
- See also: Ministry of Health (2009). Mexican Official Standard NOM-028-SSA2-2009 For the prevention, treatment and control of addictions. — http://www.conadic.salud.gob.mx/pdfs/norma_oficial_nom.pdf
- See also: World Health Organization (2005). Document of the Americas on Good Clinical Practices. Pan American Health Organization. — https://www.ms.gba.gov.ar/ssps/investigacion/DocTecnicos/BuenasPracticas-DocAmericas.pdf
- See also: World Medical Association (2013). Declaration of Helsinki. — https://www.wma.net/es/policies-post/declaracion-de-helsinki-de-la-amm-principios-eticos-para-las-investigaciones-medicas-en-seres-humanos/
- See also: World Health Organization. (2010) Global strategy to reduce the harmful use of alcohol. Geneva, Switzerland — https://pnsd.sanidad.gob.es/profesionales/publicaciones/catalogo/bibliotecaDigital/publicaciones/pdf/Organizacion_Mundial_de_la_Salud_-OMS-_(2010)_Estrategia_mundial_para_reducir_el_uso_nocivo_del_alcohol.pdf